CLINICAL TRIAL: NCT03331497
Title: Tonsillotomy or Follow-up in PFAPA -Syndrome - Randomised, Controlled Study Using Sequential Design
Brief Title: Tonsillotomy or Follow-up in PFAPA Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other); Tampere University (Other); Tampere University Hospital (Other); Turku University Hospital (Other Government); University of Turku (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TT 50_2017
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: PFAPA Syndrome
MeSH Terms: conditions — Marshall syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tonsillotomy (Experimental): The patients diagnosed with PFAPA will have tonsillotomy performed in one month from randomisation.
  Interventions: Procedure: Tonsillotomy
- Follow up (No Intervention): The patients diagnosed with PFAPA will be monitored for 3 months time. If the symptoms still persist, tonsillectomy will be performed

INTERVENTIONS:
Procedure: Tonsillotomy — About 2/3 of the palatine tonsil tissue is removed with coplator or bipolar knife.
  Arms: Tonsillotomy

SUMMARY:
Children with periodic fever, aphthous stomatitis, pharyngitis, adenitis (PFAPA) -syndrome diagnosis will be randomised either to tonsillotomy (partial tonsillectomy) or 3 months follow up. At follow up visit 3 months after randomisation the children from either groups with ongoing symptoms will be sent to tonsillectomy.

DETAILED DESCRIPTION:
Children with periodic fever, aphthous stomatitis, pharyngitis, adenitis (PFAPA) -syndrome diagnosis will be randomised either to tonsillotomy (partial tonsillectomy) or 3 months follow up.

In both groups the symptoms are monitored with symptom diaries. At follow up visit 3 months after randomisation the children from either groups with ongoing symptoms will be sent to tonsillectomy (total remove of palatine tonsil).

The design is sequential trial. From the previous trials we know that the effect of tonsillectomy is about 90% and that during follow up for six months as much as 50% of the patients will recover. Because the syndrome is rare and because the rescue operations of the tonsils (tonsillectomy in a person who has gone through tonsillotomy), the sample size has to be as low as possible. That is the reason why we chose sequential design, with assessments after every 8 patient.

Randomization is made in blocks of four. In sequential design we use the following assumptions:

* We are looking for a 40% absolute difference in cure rate between tonsillotomy (90%) and follow up (50%) groups.
* Two sided Whitehead design
* Maximum likelihood estimation (MLE)
* Five assessments (sample size 4+4, 8+8. 12+12, 16+16 and 19+19)
* type 1 error 5 % and power 80%
* The sample size will be from 8 to 38 patients depending on when the trial can be stopped along assessments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed PFAPA syndrome: regularly occurring fever episodes for 3-5 days for at least five times or for 6 months

Exclusion Criteria:

* prior tonsil surgery

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Cure | 3 months from randomization
  Proportion of patients who do not have any PFAPA symptoms

SECONDARY OUTCOMES:
Rescue surgery | 12 months from randomization
  Proportion of patients needing rescue surgery (tonsillectomy)
Days with fever | 3 months from randomization
  Number of days with fever >38C in symptom diaries
Cure | 6 months from randomization
  Proportion of patients who do not have any PFAPA symptoms

CONTACTS AND LOCATIONS:
Locations (3):
- Finland (3):
  - Oulu Unversity Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku